CLINICAL TRIAL: NCT04589689
Title: Insul-In This Together Program: Optimizing Family-based Interventions for Adolescents With Type 1 Diabetes and Their Parents
Brief Title: Insul-In This Together Program for Adolescents With Type 1 Diabetes and Their Parents
Acronym: IITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Korey Hood, Professor, Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58372; 1K23DK121771-01A1 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomization to either the intervention group (receives program immediately) or a waitlisted control condition (receives the intervention 6 months later).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will participated in the The Insul-In This Together intervention, which consists of 6 weekly 30-minute online family sessions to discuss topics related to diabetes distress and parent-teen communication. Sessions include structured education, discussions, and skill-building activities related to parental involvement, parental monitoring, and parent-adolescent conflict. The intervention will be conducted by the PI or clinically trained research staff via Zoom. Online surveys, and glucose monitoring data will be captured at baseline and 3,6 and 12-month follow-ups. Brief surveys will also be conducted at 2-, 4-, and 6-week follow-ups (after every 2 sessions for the intervention group and later the control group). Participants will be asked to provide A1C test results that will be collected via chart review or from participants sharing their test results at baseline, 6-month, and 12-month follow-up.
  Interventions: Behavioral: Insul-In This Together
- Waitlisted Control Group (Experimental): The waitlisted control group will receive the same intervention as the intervention group, but at the 6-month follow-up mark. The intervention will be conducted by the PI or clinically trained research staff via Zoom. Online surveys, and glucose monitoring data will be captured at baseline and 3,6 and 12-month follow-ups. Brief surveys will also be conducted at 2-, 4-, and 6-week from baseline. Participants will be asked to provide A1C test results that will be collected via chart review or from participants sharing their test results at baseline, 6-month, and 12-month follow-up.
  Interventions: Behavioral: Insul-In This Together

INTERVENTIONS:
Behavioral: Insul-In This Together — Session 1: Introduction to Parental Monitoring Session 2: Advanced Parental Monitoring Session 3: Introduction to Parental Involvement Session 4: Advanced Parental Involvement Session 5: Introduction to Parent-Teen Conflict Management Session 6: Advanced Parent-Teen Conflict Management

SUMMARY:
The "Insul-In This Together" intervention is designed for teens with Type 1 Diabetes and their parents. This study seeks to evaluate an evidence-based family intervention for teens with type 1 diabetes and their parents to offset the psychosocial and diabetes self-management risks. This information will provide a more in-depth understanding of family-based program efficacy for teens with adolescents and provide more judicious and streamlined intervention options to be offered in diabetes clinics in the future.

DETAILED DESCRIPTION:
This study will collect survey and biomedical data to assess this program in a randomized controlled trial with 165 families (including an adolescent and parent/caregiver) will be enrolled, complete surveys, provide biomedical data via continuous glucose monitors and receive a 6-week psychosocial intervention. The results of this study will inform future intervention redesign to provide more judicious interventions to be disseminated across diabetes care.This study will evaluate the relative efficacy of each of the individual intervention components and also identify the mechanisms of actions (mediators) that are most impacted by these types of interventions as well as most linked to long-term outcomes for adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Teen subject has a type 1 diabetes (T1D) diagnosis according to ADA criteria for at least 6 months
2. Teen subject is age 12-19 years at time of screening (no age limit for parent participants)
3. Participation of at least one cohabitating parent/caregiver.

Exclusion Criteria:

1. Subject lacks access to a smartphone or Wi-Fi via computer
2. Subject has restricted or no English proficiency
3. Subject has a pervasive developmental, cognitive, or psychiatric limitations that compromise participation in study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Korey K Hood, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was of adolescent/parent dyads, both had to sign informed consent for either of them to enroll, and they received the study intervention together.
Pre-assignment Details: 366 participants signed informed consent (representing 183 parent-adolescent dyads); 314 participants were randomized to a study arm (representing 157 adolescent-parent dyads).
Groups:
- Intervention Group - Adolescents; Intervention Group - Parents: Group assignment and intervention delivery was based on parent-adolescent dyads. The intervention group were offered the The Insul-In This Together intervention beginning immediately after baseline data collection. The intervention consists of 6 weekly 30-minute online family sessions to discuss topics related to diabetes distress and parent-teen communication, with follow-up visits through 12 months after randomization.
- Waitlisted Control Group - Adolescents; Waitlisted Control Group - Parents: Group assignment and intervention delivery was based on parent-adolescent dyads. The waitlisted control group were offered the same intervention as the intervention group, beginning after 6-month data collection completion. The intervention consists of 6 weekly 30-minute online family sessions to discuss topics related to diabetes distress and parent-teen communication, with follow-up visits through 12 months after randomization.
Period: Overall Study
Arm/Group | Intervention Group - Adolescents | Intervention Group - Parents | Waitlisted Control Group - Adolescents | Waitlisted Control Group - Parents
Started | 79 | 79 | 78 | 78
Completed | 68 | 68 | 61 | 61
Not Completed | 11 | 11 | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group - Adolescents | Intervention Group - Parents | Waitlisted Control Group - Adolescents | Waitlisted Control Group - Parents | Total
Number analyzed (Participants) | 79 | 79 | 78 | 78 | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 73 | 0 | 72 | 0 | 145
  Between 18 and 65 years | 6 | 79 | 6 | 78 | 169
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 45 | 7 | 34 | 9 | 95
  Female | 32 | 72 | 40 | 68 | 212
  Non-binary | 1 | 0 | 1 | 1 | 3
  Undisclosed | 1 | 0 | 3 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 61 | 66 | 61 | 65 | 253
  Hispanic white | 5 | 3 | 1 | 3 | 12
  Black | 2 | 1 | 3 | 2 | 8
  Asian/Pacific Islander | 2 | 4 | 2 | 7 | 15
  Native American | 0 | 1 | 0 | 0 | 1
  More than once race | 7 | 1 | 7 | 0 | 15
  Undisclosed | 2 | 3 | 4 | 1 | 10
Region of Enrollment [Count of Participants; unit: Participants] — Based on parent report and representing parent-adolescent dyads
  Participants
    United States | 79 | 79 | 78 | 78 | 314

OUTCOME MEASURES:

1. Primary Outcome: Glucose Levels Percent Time in Target Range Based on Glucose Monitoring
Description: Adolescent glucose levels percent time in target range (70-180 mg/dL) based on glucose monitoring to measure glycemic control. The clinical recommendation is a percent time-in-range of 70% or more.
Time Frame: Average percent time in range based on two weeks of glucose monitoring data at baseline, 3-month, and 6-month follow-up (plus or minus 2 weeks around target data collection date)
Population: Enrolled adolescents; data for this outcome were not collected from parents
Measure: Mean (Standard Deviation); unit: percentage of time-in-range
Groups:
- Intervention Group: The intervention group were offered the The Insul-In This Together intervention beginning immediately after baseline data collection. The intervention consists of 6 weekly 30-minute online family sessions to discuss topics related to diabetes distress and parent-teen communication, with follow-up visits through 12 months after randomization.
- Waitlisted Control Group: The waitlisted control group were offered the same intervention as the intervention group, beginning after 6-month data collection completion. The intervention consists of 6 weekly 30-minute online family sessions to discuss topics related to diabetes distress and parent-teen communication, with follow-up visits through 12 months after randomization.
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
percentage of time-in-range
  Baseline | 61.185 (18.42) | 64.542 (17.74)
  3 months | 62.223 (18.57) | 64.571 (18.21)
  6 months | 61.680 (18.91) | 65.908 (17.82)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3 months; Test type: Other; p = 0.777, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month; Test type: Other; p = 0.247, t-test, 2 sided — The a priori threshold for statistical significance is <.05

2. Primary Outcome: Adolescent Quality of Life
Description: Self-report via Type 1 Diabetes and Life (T1DAL) surveys for adolescents to measure the adolescent's quality of life. Possible score range is 0-100 and the higher scores indicated better quality of life. Adolescent quality of life was measured for adolescents only (not parents).
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up.
Population: Enrolled adolescents; data for this outcome were not collected from parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 67.902 (13.92) | 64.633 (15.38)
  3-month | 67.965 (14.47) | 63.675 (16.39)
  6-month | 69.523 (14.63) | 65.511 (16.16)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.160, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.275, t-test, 2 sided — The a priori threshold for statistical significance is <.05

3. Secondary Outcome: Adolescent Depression
Description: Surveys of self-report via Children's Depression Inventory - short version (CDI:S80), a 10 scale item, will be used to assess adolescent depression. Possible total score range is 0-20 with higher scores indicated more severe depressive symptoms. Item response options included 0 = Not at all, 1 = Somewhat, and 2 = A lot. Total score was the sum of all item scores.
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up.
Population: Enrolled adolescents; data for this outcome were not collected from parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 2.278 (3.56) | 2.718 (3.63)
  3-month follow-up | 2.411 (4.27) | 3.130 (3.91)
  6-month follow-up | 2.419 (4.01) | 2.963 (3.96)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.509, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.610, t-test, 2 sided — The a priori threshold for statistical significance is <.05

4. Secondary Outcome: Parent Depression
Description: Surveys of self-report via the Patient Health Questionnaire (PHQ-8) - 8 item scale to assess depression among parents. Response options for each item included 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day. Items were summed into a total score. The possible total score range is 0-24 and higher scores indicate more depressive symptoms.
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up.
Population: Enrolled parents; data for this outcome were not collected from adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 4.772 (4.82) | 5.167 (5.25)
  3-month follow-up | 4.099 (4.02) | 4.346 (4.81)
  6-month follow-up | 4.088 (4.56) | 4.409 (4.43)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.807, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.826, t-test, 2 sided — The a priori threshold for statistical significance is <.05

5. Secondary Outcome: Adolescent Diabetes Distress
Description: Measured by the Problem Areas In Diabetes (PAID) survey of diabetes distress, which includes 14 items that were summed to create a total score with a possible total score range of 14-84. Item response options range from 1 (not a problem) to 6 (serious problem). Higher scores indicate more diabetes distress.
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up
Population: Enrolled adolescents; data for this outcome were not collected from parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 28.608 (12.68) | 32.064 (14.98)
  3-month follow-up | 27.847 (13.07) | 32.219 (16.39)
  6-month follow-up | 27.883 (11.97) | 30.265 (16.16)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.076, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.747, t-test, 2 sided — The a priori threshold for statistical significance is <.05

6. Secondary Outcome: Parent Diabetes Distress
Description: Measured by the Problem Areas In Diabetes (PAID) survey of diabetes distress, which includes 15 items that were summed into a total score with a possible total score range of 15-90. Higher scores indicate more diabetes distress. Response options ranged from 1 (not a problem) to 6 (serious problem).
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up.
Population: Enrolled parents; data for this outcome were not collected from adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 43.177 (17.32) | 44.859 (17.81)
  3-month follow-up | 36.405 (14.27) | 38.817 (16.22)
  6-month follow-up | 36.393 (14.39) | 40.542 (18.09)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.154, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.107, t-test, 2 sided — The a priori threshold for statistical significance is <.05

7. Secondary Outcome: Parenting Stress
Description: Surveys of self-report on parenting stress via The Parenting Stress Scale. Includes 18 items that were summed into a total score with a possible total score range from 18-90. Higher scores indicate more parenting stress. Item responses included 1 = strongly agree, 2 = agree, 3 = not sure, 4 = disagree, and 5 = strongly disagree.
Time Frame: Baseline, 3-month follow-up, and 6-month follow-up
Population: Enrolled parents; data for this outcome were not collected from adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 79 | 78
score on a scale
  Baseline | 73.633 (9.73) | 71.256 (10.88)
  3-month follow-up | 74.706 (9.16) | 71.777 (12.25)
  6-month follow-up | 74.376 (9.73) | 71.865 (10.93)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 3-month follow-up; Test type: Other; p = 0.445, t-test, 2 sided — The a priori threshold for statistical significance is <.05
Statistical Analysis 2: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.543, t-test, 2 sided — The a priori threshold for statistical significance is <.05

8. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Medical record data on glycated hemoglobin in blood reported as National Glycohemoglobin Standardization Program (NGSP) percentage. The clinical recommendation for pediatrics is below 7.5%.
Time Frame: Baseline and 6-month follow-up
Population: Enrolled adolescents with available data; data for this outcome were not collected from parents
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention Group | Waitlisted Control Group
Number analyzed (Participants) | 77 | 75
percentage of glycated hemoglobin
  Baseline | 7.166 (1.20) | 7.19 (1.42)
  6-month follow-up | 7.260 (1.38) | 7.069 (1.29)
Statistical Analysis 1: Comparison: Intervention Group vs Waitlisted Control Group; Analysis at 6-month follow-up; Test type: Other; p = 0.157, t-test, 2 sided — The a priori threshold for statistical significance is <.05

ADVERSE EVENTS:
Time Frame: Up to 12 months
Groups:
- Intervention Group - Adolescents: Data for adolescents in the dyads of the intervention group during their intervention period.
- Intervention Group - Parents: Data for parents in the dyads of the intervention group during their intervention period.
- Waitlisted Control Group: Control - Adolescents: Data for adolescents in the dyads of the waitlisted group during their waiting (control) period.
- Waitlisted Control Group: Control - Parents: Data for parents in the dyads of the waitlisted group during their waiting (control) period.
- Waitlisted Control Group: Intervention - Adolescents: Data for adolescents in the dyads of the waitlisted group during their intervention period.
- Waitlisted Control Group: Intervention - Parents: Data for parents in the dyads of the waitlisted group during their intervention period.
Arm/Group | Intervention Group - Adolescents | Intervention Group - Parents | Waitlisted Control Group: Control - Adolescents | Waitlisted Control Group: Control - Parents | Waitlisted Control Group: Intervention - Adolescents | Waitlisted Control Group: Intervention - Parents
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/79 | 0/78 | 0/78 | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/78 | 0/78 | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/78 | 0/78 | 0/78 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04589689/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04589689/SAP_001.pdf